CLINICAL TRIAL: NCT02979678
Title: The Update of the EORTC Quality of Life Questionnaire Breast Cancer Module (EORTC QLQ-Breast 23) Phase 1-3
Brief Title: European Organisation of Research and Treatment (EORTC) Quality of Life Questionnaire (QLQ) Breast Cancer Module Update
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 27-355
Record Dates: First submitted 2016-10-13; First posted 2016-12-01 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Quality of Life
Keywords: Breast cancer, quality of life
MeSH Terms: conditions — Breast Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Questionnaire (Experimental): Breast cancer
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — The questionnaire should be updated with respect to wording, terminology.
  Other Names: EORTC QLQ-Breast Cancer Module Update

SUMMARY:
The purpose of this study is to update the EORTC QLQ Breast (BR)-23 Module. Since the development of BR-23 published 1996 the standard therapy of breast cancer has changed. New therapies brought new side effects and different impact on QoL (quality of life) are not sufficiently covered by EORTC QLQ BR-23 and an update of the module could be useful, both from clinical and scientific point of view.

DETAILED DESCRIPTION:
1. Based on a systematic literature search a new issue list will be developed, containing additional issues relevant for new treatment strategies. A total of 5-10 patients from different countries (5-8) as well as health care professionals (5/country) will be interviewed (Phase 1).
2. Operationalization of the issues into items; a provisional version of a the questionnaire and a hypothetic scale structure will be established (Phase2).
3. The resulting provisional updated module will be tested with respect to understanding, comprehensiveness and applicability (according to the EORTC Module Development Guidelines). The items will be translated from English into other languages following a standardized forward-backward procedure. Total aof 260 patients will be interviewed from different cultural areas: Northern Europe, Central Europe, Southern Europe, Asia (Phase 3).
4. The module and its scale structure will be field-tested in a large, international group of patients in order to determine its acceptability, reliability, validity, responsiveness and crosscultural applicability .

ELIGIBILITY:
Inclusion Criteria:

* Patients with early or metastatic breast cancer

Exclusion Criteria:

* Patients with second malignancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2015-06; Primary Completion 2018-03 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Quality of life | 3 years, Patients under treatment are asked once to complete the questionnaire during 3 years
  Patients under Treatment are asked to complete the questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Vesna Bjelic-Radisic, Principal Investigator — Medical University of Graz
Locations (9):
- Medical University Graz, Graz, Austria
- University Hospital Centre Rijeka, Rijeka, Croatia
- Institut de Cancerologie de Lorraine, Lorraine, France
- University Medical Center Regensburg, Regensburg, Germany
- Italy (2):
  - Instituto Nazionale Tumori Fondazione Pascale, Naples
  - IOV Oncologico Veneto Padova, Padivarma
- Netherlands Cancer Institute - NKI, Amsterdam, Netherlands
- Jagiellonian University Medical College Krakow, Krakow, Poland
- Oncology Department Hospital of Navarre, Navarra, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sprangers MA, Groenvold M, Arraras JI, Franklin J, te Velde A, Muller M, Franzini L, Williams A, de Haes HC, Hopwood P, Cull A, Aaronson NK. The European Organization for Research and Treatment of Cancer breast cancer-specific quality-of-life questionnaire module: first results from a three-country field study. J Clin Oncol. 1996 Oct;14(10):2756-68. doi: 10.1200/JCO.1996.14.10.2756. PMID 8874337
- [Result] Johnson C, Aaronson N, Blazeby JM et al. Guidelines for Developing Questionnaire Modules. 4ed.Bruessels, EORTC,2011